CLINICAL TRIAL: NCT03141827
Title: The Effect of Intranasal Insulin on Hepatic and Intestinal Triglyceride-rich Lipoprotein Production
Acronym: LPNI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: LPNI-REB-15-9475
Record Dates: First submitted 2017-05-03; First posted 2017-05-05 (Actual); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Hyperlipidemia
Keywords: Lipoprotein; Apolipoprotein; Pancreatic clamp; Insulin; Nasal
MeSH Terms: conditions — Hyperlipidemias; Insulin Resistance | interventions — Insulin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin (Experimental): Nasal spray, insulin 40 IU, single dose
  Interventions: Drug: Insulin
- Placebo (Placebo Comparator): Nasal spray, placebo, single dose
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Insulin — Insulin 40 IU, nasal spray, single dose
  Arms: Insulin
Drug: Placebo — Placebo, nasal spray, single dose
  Arms: Placebo

SUMMARY:
This study compares the effect of insulin given as a nasal spray with a placebo. Insulin is a chemical messenger (hormone) in the body that controls fat (triglyceride) levels in the blood by controlling the amount of fat made by the liver and gut. Recent research suggests that insulin may work through the brain. The investigators hypothesize that preferential delivery of insulin into the brain, through nasal spray of the hormone, may affect the amount of fats made by the liver and gut.

DETAILED DESCRIPTION:
Each subject will be studied twice 4-6 weeks apart in random order in this single blinded study. In study A they will receive a single dose of insulin 40 IU through nasal spray. In study B they will receive placebo. On the day of the study subjects will drink regular liquid nutrient formula to maintain a constant fed state. A pancreatic clamp (octreotide with replacement glucose, insulin and growth hormone) will be started at 7am. From 9am a regular infusion of a stable isotope tracer will be started together with nasal spray of either insulin/placebo. Regular blood samples will be drawn to assess lipoprotein kinetics.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, aged 18 to 60 years
2. Body mass index 20 to 40 kg/m2
3. Hemoglobin in the normal range.
4. Normal glucose tolerance in response to a 75g, 2-hr oral glucose tolerance test
5. Women of reproductive age should be on contraception (oral contraceptive pill or intra-uterine device/coil) for at least 2 months prior to and after the study.

Exclusion Criteria:

1. Study participant with a history of hepatitis/hepatic disease that has been active within the previous two years.
2. Any current or previous history of biliary disease (including gall stones, biliary atresia and cholecystitis) or pancreatitis.
3. Any current or previous history of endocrine disease, dyslipidemia or malignancy
4. Any significant active (over the past 12 months) disease of the gastrointestinal, pulmonary, neurological, renal (creatinine > 1.5 mg/dL) genitourinary, hematological systems, or has severe uncontrolled treated or untreated hyper/ hypotension (sitting diastolic pressure > 100 or systolic > 180 or systolic pressure <100) or proliferative retinopathy
5. Use of immunosuppressive agents at any time during the study
6. Allergy to any study medication
7. Pregnancy or breastfeeding
8. Heavy smoker
9. Fasting blood glucose > 6.0 mmol/l or known diabetes.
10. Any history of a myocardial infarction or clinically significant, active, cardiovascular history including a history of arrhythmia's or conduction delays on electrocardiogram, unstable angina, or decompensated heart failure.
11. Any nasal pathology.
12. Any laboratory values: aspartate aminotransferase > 2x upper limit of normal ; alanine aminotransferase > 2x upper limit of normal; thyroid-stimulating hormone > 6 milliunit per litre

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2016-04-14 (Actual); Primary Completion 2017-02-15 (Actual); Study Completion 2017-04-26 (Actual)

PRIMARY OUTCOMES:
Triglyceride-rich lipoprotein apolipoprotein B100 production rate | 10 hours
  Triglyceride-rich lipoprotein apolipoprotein B100 production rate will be measured following nasal spray of insulin or placebo

SECONDARY OUTCOMES:
Triglyceride-rich lipoprotein apolipoprotein B48 production rate | 10 hours
  Triglyceride-rich lipoprotein apolipoprotein B48 production rate will be measured following nasal spray of insulin or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Gary F Lewis, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Tornto General Hospital, UHN, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Xiao C, Dash S, Stahel P, Lewis GF. Effects of Intranasal Insulin on Triglyceride-Rich Lipoprotein Particle Production in Healthy Men. Arterioscler Thromb Vasc Biol. 2017 Sep;37(9):1776-1781. doi: 10.1161/ATVBAHA.117.309705. Epub 2017 Jul 27. PMID 28751575